CLINICAL TRIAL: NCT02668744
Title: Texas Sprouts: A School-based Gardening Obesity Intervention for Low-income Minority Children
Brief Title: A School-based Gardening Obesity Intervention for Low-income Minority Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); The University of Texas Health Science Center, Houston (Other); Seton Healthcare Family (Other); Texas AgriLife Extension Service (Other)
Responsible Party: Principal Investigator, Jaimie N. Davis, Associate Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01HL123865-01A1 (NIH); R01HL123865 (NIH)
Record Dates: First submitted 2016-01-19; First posted 2016-01-29 (Estimated); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): TX Sprouts
  Interventions: Behavioral: Intervention
- Control (Placebo Comparator): Delayed Intervention
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — The intervention consists of building edible gardens at each the eight participating and eligible schools. Educators will be provided to lead 18 gardening, nutrition and cooking lessons throughout the school year intervention to all 3-5th grade students. Nine gardening, nutrition, and cooking classes will be taught to parents every month. Garden Leadership Coalitions (GLCs), made up of parents, teachers and school staff, will be formed and training/resources provided to help with adoption of the program. Training and resources will be provided to the GLCs and teachers in the 2nd year to assist with sustainability.

SUMMARY:
The investigators recently completed an NIH R21 grant, which was a randomized controlled trial (RCT) to test the effects of a gardening, nutrition, and cooking program in 375 low-income Hispanic students living in Los Angeles. Preliminary results from this study show that intervention compared to the control students have reductions in BMI parameters and waist circumference, increases in daily intake of dietary fiber and vegetables, and improved lipid profiles. The investigators want to expand and replicate this study by: a) using a cluster randomized school design; b) implementing the program during school hours; c) increasing sample size; d) lengthening the intervention period to one school year; e) collecting comprehensive metabolic measurements on the child; f) enhancing family workshops; g) collecting more parental data; and h) developing and evaluating sustainability strategies. Thus, the overall goal of this project is to test the effects of a large school-based gardening, nutrition, and cooking RCT (called "Sprouts") on dietary intake, dietary-related behaviors, obesity, and related metabolic disorders in low-income Hispanic youth and their families in Central Texas. Sixteen elementary schools will be randomized to either: 1) Sprouts intervention or 2) Control (delayed intervention). At each intervention school, the investigators will build edible gardens; form and train Garden Leadership Coalitions (GLCs); teach 20 Sprouts in-school lessons to the students; and teach nine family-based Sprouts lessons throughout school year. The following measures will be obtained for students at baseline and post-intervention: height, weight, BMI, waist circumference, body composition (via bioimpedance), blood pressure, glucose, insulin, and lipids (via voluntary fasting blood draws), dietary intake, and related psychosocial behaviors (e.g., preference/motivation/self-efficacy to eat FV). The investigators will also measure anthropometrics, dietary intake, and related dietary psychosocial variables on the parents at baseline and post-intervention. After the intervention year, the investigators will provide a series of training workshops and resources to the GLCs and schoolteachers to sustain the Sprouts program in subsequent years. The investigators will measure the sustainability employed by each school by process logs/surveys, structured interviews, and school observations.

DETAILED DESCRIPTION:
Garden Leadership Coalition (GLC): The investigators will establish GLCs at each of the schools during the intervention phase, which will facilitate some of the school-level components of the intervention. These GLCs will be comprised of interested teachers, school staff, senior citizens, parents, and children, but these groups will be different and unique at each school site.

Edible Gardens: Raised beds will be used at all garden sites, as these are easy to build, make garden access easy for children of all developmental levels, ensure that soils are free of heavy metals/contaminants, and reduce weeds in the garden area. Each school site will get the materials and supplies needed for garden upkeep and for teaching the lessons,.

Curriculum: A total of 18 lessons (1 hour each) will be taught weekly over the course of the intervention year. The curriculum is culturally tailored to Hispanics, including culturally appropriate recipes, content, and activities. The curriculum is mapped on State of Texas Assessments of Academic Readiness (STAAR) standards for science, math, language arts, health, and social studies. The 9 parent lessons (each 1 hour long) will parallel the nutrition and gardening topics/activities taught to the children. The parent curriculum is available in both English and Spanish and has been culturally adapted and evaluated. The curriculum has a strong emphasis on the cooking components and focuses on growing and cooking foods that are culturally appropriate.

School Lessons: The investigators will hire bilingual nutrition and garden educators who have experience teaching nutrition/ gardening programs to teach the Sprouts curriculum. Lessons will be taught by our educators separately to each 3rd-5th grade classroom throughout the school year as part of their normal school day. Although nutrition and garden educators will be provided to teach these lessons the first year, the schoolteachers will attend all of these lessons, providing the initial training for them to continue the program in subsequent years.

Family Lessons at Schools: The bilingual garden/nutrition educators will also teach monthly Sprouts lessons throughout the school year for the families of participants at each of the schools.

Delayed Intervention to Control Schools: The control schools will receive a delayed intervention (identical intervention as described above) in the year after the post-testing for that wave. Baseline and post-intervention measurements will occur in the control parents and students within the same time period as the intervention schools. Every control school will receive a garden, identical in size and structure to the intervention schools.

Evaluation Measures: Evaluation measures will be collected at baseline and end of the school year in both arms (intervention and control schools). Measurements will occur during the first four weeks of school in the fall and the last four weeks of school in the spring. Most measures on children will be collected at the schools during normal school hours, whereas the blood draw will be collected on school campuses before school starts. Parent questionnaires will be handed out or mailed to the homes after consent is obtained. The questionnaires are translated into Spanish, culturally appropriate, and take ~60 minutes to complete.

Anthropometrics, Body Fat, and Blood Pressure: For both children and parents, weight will be measured using a digital scale to the nearest 0.1 kg, and height will be measured using a wall-mounted stadiometer to the nearest 0.1 cm. BMI (kg/m2) and BMI percentiles for the Center for Disease Control (CDC) age- and gender-specific values will be used. Waist circumferences (WC) will be measured and recorded to the nearest 0.1 cm. Body composition will be assessed using Bioelectrical Impedance with the Tanita Body Fat Analyzer. Blood pressure will be obtained in duplicate with an automatic cuff according to recommendations of the American Heart Association. Parental height, weight, body fat, WC, and blood pressure will be collected at first and last family workshop (expecting a subsample only). Therefore the investigators will ask self-reported height and weight in questionnaire packets.

Dietary Intake: The questionnaire will use the School Physical Activity and Nutrition Project diet intake questions, which was designed to assess children's intake by food group, with a specific focus on fruit and fruit juices, vegetables, potatoes (including and excluding French fries), whole grains, meat/poultry/fish, dairy, legumes, saturated fat, and "added sugars" (in sweetened cereals, soft drinks, and sweets). The investigators will also collect 24-hour diet recalls in a subset of children. Trained interviewers will collect three recalls by telephone. All recall data will be analyzed using the Nutrition Data System for Research (NDS-R 2012, University of Minnesota).

Demographic and Dietary Psychosocial Measures: Demographic information including age, socioeconomic status and ethnicity will be obtained via a questionnaire. Parents will fill out a brief medical history form for their child and themselves to rule out exclusion criteria. Children and parents will complete questionnaires to assess preference and motivation for fruit and vegetable Intake, self-efficacy to garden, cook, and eat FV, food insecurities, and home eating environment. All parent questionnaires will be available in both English and Spanish, and written at a 3rd grade reading level.

Fasting Blood Sample: Certified phlebotomists will perform the fasting blood draws on students first thing in the morning before school starts at the schools at baseline and at the end of the school year. Students with parental consent and assent will participate in the blood draw. Students who do not assent to participate in the blood draw will still be allowed to participate in the Sprouts program. Fasting blood will be drawn to assess glucose, insulin, lipids, and adipocytokines. Blood samples will be spun, aliquoted, frozen, and transported to the University of Texas (UT) campus for assaying. All children with elevated glucose levels (in the abnormal or Type 2 diabetes range) or elevated blood pressure will be contacted via telephone by Dr. Pont (Co-I on this study) to explain the test results and be referred immediately to a health clinic for follow-up. However, these children will still be allowed to participate in the study.

Train the Trainer Workshops: At the beginning of the sustainability year, our educators will lead three "train the trainer" workshops. Schoolteachers will be given complete curriculum manuals, electronic copies of all student curriculum, and have access to all teaching material needed for every lesson. The workshops will connect teachers to community resources and will train the teachers in: structure/flow of lessons, all lesson activities/content, cooking/preparation skills, and available resources/materials.

Sustainability Measures: During the Sprouts intervention and sustainability year, the investigators will collect pilot data on sustainability strategies being implemented in both the intervention and control schools. Structured interviews will be conducted with GLC members to document member information, leadership structure, meeting times/places, how the garden was designed/built, workshops offered/attended, fundraising and media events, types of produce harvested, produce use and distribution plans, community resources leveraged, barriers and future action plans. Structured interviews will be conducted with teachers, principals, administration staff, GLCs, and district directors and staff to evaluate various aspects of the program including: a) use and maintenance of garden; b) successful and unsuccessful components/strategies implemented to sustain program; and c) additional material/resources/training requested and/or needed.

Participant Screening/Recruitment: Sixteen elementary schools will be allocated to either Sprouts intervention (n=8 schools) or Control group (n=8 schools). All participants and their parents will have to sign assent and consent forms, approved by UT-Austin's Institutional Review Board. Based on previous intervention work with Hispanic communities, the investigators anticipate ~50% of parents will consent for their children to participate, and their children will complete all the baseline measures. The investigators anticipate 15% attrition at post-intervention measurement due to parents/students moving away or being sick or absent from school. Based on parental participation rates in Los Angeles (LA) Sprouts, the investigators anticipate that 25% of parents will return parental baseline questionnaires, and the investigators assume a 15% attrition rate at post-testing. Based on blood draw participation rates in LA Sprouts, the investigators anticipate that 50% of participating children (n=1,200) will also participate in the blood draws at pre-intervention and 40% (n=960 or 60 per school) at post-intervention.

Data Management and Analyses: Data will be merged, edited, and cleaned using system files created with REDCap (Research Electronic Data Capture), which is a secure web application for building and managing databases. The database is ideal for field data collection and will be accessible to all key personnel at any location. All data will be entered using the double data entry method.

Summary statistics, graphical analyses, and frequency distributions will be used to describe the data between the intervention and control groups. Data will be transformed if needed. The investigators will handle missing data using two primary approaches: multiple imputation and full information maximum likelihood estimation methods. For Aim 1: The investigators will test if the children and parents participating in Sprouts compared to control will have increased changes in average consumption of vegetable servings per day and decreased average changes in BMI z-scores, waist circumference, fasting glucose, and insulin using well-known statistical methods for cluster randomized trials. Several analytic strategies will be employed to determine the effect of the intervention on vegetable intake and many of the other primary outcome variables. The investigators plan to conduct a two-stage nested analysis of variance model, which is a special case of the mixed effects linear regression model also known as a repeated measures analysis of variance model. The terms in the model include the true mean for the outcome variable, the fixed effects of the intervention arm, one random cluster effect (school), and the random error term. In this case, the schools (clusters) should be regarded as nested within the intervention arms and the students or parents within the school (clusters). The analytic approach for the secondary outcome measures (i.e., blood pressure, percent body fat, metabolic syndrome, adipocytokines, other dietary intake variables, and related dietary psychosocial behaviors) will involve a similar use of linear mixed models. For Aim 2: To test the effects of the Sprouts intervention on changes in vegetable intake and availability and on related dietary behaviors in the parents, the investigators will use similar and well-known statistical methods as described for Aim 1. For the Exploratory Aim, the investigators will conduct descriptive statistics on the collected pilot data of the sustainability strategies (qualitative and quantitative data obtained via structured interviews and focus groups) on both intervention and control schools.

ELIGIBILITY:
Inclusion Criteria:

* Weight status: Normal weight children (age- and sex-specific BMI<85th percentile based on CDC BMI growth charts68) and overweight and obese children (BMI≥85th percentile).
* Gender and Age: Students in 3rd-5th grades (8 to 11 y) and their parents
* Hispanic Origin: This study will include all ethnicities/races; however, the selected schools are >50% Hispanic, and therefore, we expect the majority of our students and parents to be Hispanic.

Exclusion Criteria:

* Children or parents presently taking medication(s) or diagnosed with any disease that could influence dietary intake or body composition
* Previously diagnosed with any major illness since birth (e.g. chronic birth asphyxia, cancer, etc.)
* Any physical, cognitive, or psychological disability that would prevent participation in the study.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3302 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
To test the effect of the Sprouts intervention on the changes in dietary intake (fruit and vegetables servings) in the children. | One year
  Evaluation measures will be collected one time at baseline and end of the school year in both arms (intervention and control schools). A child questionnaire will be administered and include questions about dietary intake of fruits and vegetables to assess their eating habits.
To test the effect of the Sprouts intervention on the changes in BMI in the children. | One year
  Evaluation measures will be collected one time at baseline and end of the school year in both arms (intervention and control schools). Measurements will occur during the first four weeks of school in the fall and the last four weeks of school in the spring.
  Weight will be measured using a SECA (model 869) digital scale to the nearest 0.1 kg, and height will be measured using a wall-mounted stadiometer to the nearest 0.1 cm. BMI (kg/m2) and BMI percentiles for CDC age- and gender-specific values will be determined using EpiInfo 2005.

SECONDARY OUTCOMES:
To test the effect of the Sprouts intervention on the changes in dietary intake (fruit and vegetables servings) in the parents. | One year
  Evaluation measures will be collected one time at baseline and end of the school year in both arms (intervention and control schools). A parent questionnaire will be administered and include questions about dietary intake of fruits and vegetables to assess their eating habits.
To test the effect of the Sprouts intervention on changes in BMI in the parents. | 4 years
  Evaluation measures will be collected one time at baseline and end of the school year in both arms (intervention and control schools). Measurements will occur during the first four weeks of school in the fall and the last four weeks of school in the spring.
  Weight will be measured using a SECA (model 869) digital scale to the nearest 0.1 kg, and height will be measured using a wall-mounted stadiometer to the nearest 0.1 cm. BMI (kg/m2) and BMI percentiles for CDC age- and gender-specific values will be determined using EpiInfo 2005.

CONTACTS AND LOCATIONS:
Overall Officials: Jaimie N Davis, PhD, Principal Investigator — University of Texas at Austin
Locations (16):
- United States (16):
  - Barbara Jordan Elementary, Austin, Texas
  - Decker Elementary, Austin, Texas
  - Oak Meadows Elementary, Austin, Texas
  - Pleasant Hill Elementary, Austin, Texas
  - Casey Elementary, Austin, Texas
  - Hart Elementary, Austin, Texas
  - McBee Elementary, Austin, Texas
  - Booker T. Washington, Elgin, Texas
  - Elgin Elementary, Elgin, Texas
  - Neidig Elementary, Elgin, Texas
  - Carver Elementary, Georgetown, Texas
  - Mitchell Elementary, Georgetown, Texas
  - Pickett Elementary, Georgetown, Texas
  - Purl Elementary, Georgetown, Texas
  - Callison Elementary, Round Rock, Texas
  - Voigt Elementary, Round Rock, Texas

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared. Only aggregate data.

REFERENCES:
- [Derived] Haushalter K, Burgermaster M, Hudson E, Landry MJ, Sharma SV, Davis JN. An Increase in Food Insecurity Correlated with an Increase in Plasma Triglycerides among Latinx Children. J Nutr. 2024 Feb;154(2):565-573. doi: 10.1016/j.tjnut.2023.12.024. Epub 2023 Dec 17. PMID 38110183
- [Derived] Jeans MR, Landry MJ, Vandyousefi S, Hudson EA, Burgermaster M, Bray MS, Chandra J, Davis JN. Effects of a School-Based Gardening, Cooking, and Nutrition Cluster Randomized Controlled Trial on Unprocessed and Ultra-Processed Food Consumption. J Nutr. 2023 Jul;153(7):2073-2084. doi: 10.1016/j.tjnut.2023.04.013. Epub 2023 Apr 26. PMID 37116658
- [Derived] Vandyousefi S, Ranjit N, Landry MJ, Jeans M, Ghaddar R, Davis JN. Dietary Psychosocial Mediators of Vegetable Intake in Schoolchildren From Low-Income and Racial and Ethnic Minority US Families: Findings From the Texas Sprouts Intervention. J Acad Nutr Diet. 2023 Aug;123(8):1187-1196.e1. doi: 10.1016/j.jand.2023.03.015. Epub 2023 Mar 28. PMID 36996935
- [Derived] Davis JN, Landry MJ, Vandyousefi S, Jeans MR, Hudson EA, Hoelscher DM, van den Berg AE, Perez A. Effects of a School-Based Nutrition, Gardening, and Cooking Intervention on Metabolic Parameters in High-risk Youth: A Secondary Analysis of a Cluster Randomized Clinical Trial. JAMA Netw Open. 2023 Jan 3;6(1):e2250375. doi: 10.1001/jamanetworkopen.2022.50375. PMID 36626172
- [Derived] Jeans MR, Ghaddar R, Vandyousefi S, Landry MJ, Gray MJ, Leidy HJ, Whittaker TA, Bray MS, Davis JN. Distinct racial and ethnic metabolic syndrome characteristics: A comparative assessment in low-income children 7-10 years of age. Pediatr Obes. 2022 Oct;17(10):e12925. doi: 10.1111/ijpo.12925. Epub 2022 May 12. PMID 35560860
- [Derived] Jeans MR, Landry MJ, Asigbee FM, Vandyousefi S, Ghaddar R, Bray MS, Leidy HJ, Davis JN. Comparison of School vs Home Breakfast Consumption with Cardiometabolic and Dietary Parameters in Low-Income, Multiracial/Ethnic Elementary School-Aged Children. J Acad Nutr Diet. 2022 Apr;122(4):833-847. doi: 10.1016/j.jand.2021.10.014. Epub 2021 Oct 9. PMID 34634512
- [Derived] Landry MJ, van den Berg AE, Hoelscher DM, Asigbee FM, Vandyousefi S, Ghaddar R, Jeans MR, Waugh L, Nikah K, Sharma SV, Davis JN. Impact of a School-Based Gardening, Cooking, Nutrition Intervention on Diet Intake and Quality: The TX Sprouts Randomized Controlled Trial. Nutrients. 2021 Sep 1;13(9):3081. doi: 10.3390/nu13093081. PMID 34578959
- [Derived] Davis JN, Perez A, Asigbee FM, Landry MJ, Vandyousefi S, Ghaddar R, Hoover A, Jeans M, Nikah K, Fischer B, Pont SJ, Richards D, Hoelscher DM, Van Den Berg AE. School-based gardening, cooking and nutrition intervention increased vegetable intake but did not reduce BMI: Texas sprouts - a cluster randomized controlled trial. Int J Behav Nutr Phys Act. 2021 Jan 23;18(1):18. doi: 10.1186/s12966-021-01087-x. PMID 33485354
- [Derived] Landry MJ, van den Berg AE, Asigbee FM, Vandyousefi S, Ghaddar R, Davis JN. Child Compared with Parent Perceptions of Child-Level Food Security. Curr Dev Nutr. 2019 Sep 27;3(10):nzz106. doi: 10.1093/cdn/nzz106. eCollection 2019 Oct. PMID 31637366
- [Derived] Landry MJ, Ranjit N, Hoelscher DM, Asigbee FM, Vandyousefi S, Ghaddar R, Davis JN. Validity and Reliability of an Expanded Vegetable Questionnaire Among Elementary School Children. Curr Dev Nutr. 2019 Jul 4;3(8):nzz080. doi: 10.1093/cdn/nzz080. eCollection 2019 Aug. PMID 31414072